CLINICAL TRIAL: NCT04985279
Title: Position and Angle Marking System (PAMS) for Ultrasound-guided Neuraxial Procedures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: KK Women's and Children's Hospital (Other Government)
Responsible Party: Principal Investigator, Paul Tan Hon Sen, Associate Consultant, KK Women's and Children's Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PAMS 2021/2159
Record Dates: First submitted 2021-07-05; First posted 2021-08-02 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Ultrasound-guided Neuraxial Procedures
Keywords: Ultrasonography; Epidural; Spinal; Labour analgesia
MeSH Terms: interventions — Patient Positioning

STUDY DESIGN:
Intervention Model Description: The ultrasound operators will be randomised to perform either
  1. Skin marking after lumbar ultrasonography using marker pens (standard practice)
  2. Skin marking after lumbar ultrasonography using PAMS
  After completion of the first procedure, the ultrasound operators will then crossover and perform the other procedure.
Masking Description: No masking involved.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard clinical practice (Active Comparator): * Lumbar ultrasound scan will be performed to identify the desired needle insertion site, followed by demarcation using skin markers.
  * The angulation of the ultrasound probe will be adjusted to optimise the image of the simulated patient's lumbar spine.
  * The ultrasound probe will be removed and needle insertion simulated by touching the tip of a blunt needle to the patient's back, at the desired angle.
  * A usability questionnaire regarding the procedure will be completed.
  Interventions: Device: Standard clinical practice
- Position and Angle Marking System (PAMS) (Experimental): * PAMS will be attached to the ultrasound probe.
  * Lumbar ultrasound scan will be performed to identify the desired needle insertion site, followed by demarcation by gentle pressing PAMS into the simulated patient's back to create skin indentations.
  * The angulation of the ultrasound probe will be adjusted to optimise the image of the simulated patient's lumbar spine, and the angle read off a graduated scale.
  * The ultrasound probe will be removed and needle insertion simulated by touching the tip of a blunt needle to the patient's back, at the desired angle.
  * A usability questionnaire regarding the procedure will be completed.
  Interventions: Device: Position and Angle Marking System

INTERVENTIONS:
Device: Position and Angle Marking System — Position and Angular Marking System (PAMS) attaches on to the ultrasound probe. When the desired insertion site is identified by ultrasound, the doctor gently presses PAMS into the patient's back to create skin indentations demarcating the needle insertion point. These indentations are not affected by skin sterilisation, and may improve accuracy and reduce the time taken to perform the epidural procedure. Next, the angle between the ultrasound probe and the patient's back can be measured using PAMS, and this angle can be maintained using a needle guide during the epidural procedure.
  Other Names: PAMS
  Arms: Position and Angle Marking System (PAMS)
Device: Standard clinical practice — When the desired insertion site is identified by ultrasound, the doctor demarcate the needle insertion point using marker pens.
  Arms: Standard clinical practice

SUMMARY:
Epidural anaesthesia involves the administration of numbing medication (local anaesthetics) close to the spinal canal, and is regarded as the best method for providing pain relief during labour and childbirth. The use of ultrasound to guide epidural insertion and placement has been shown to improve pain relief and reduce the risk of complications.

However, after identifying the desired needle insertion site via ultrasound, current practice involves demarcating the insertion site using marker pens, which is time-consuming, inaccurate, and may be inadvertently removed by skin sterilisation. Furthermore, the desired needle angulation determined by ultrasound cannot be accurately measured and maintained during the epidural procedure. Both issues limit the benefits of using ultrasound to guide the epidural procedure.

To address these issues, the investigators developed a Position and Angular Marking System (PAMS) that attaches on to the ultrasound probe. When the desired insertion site is identified by ultrasound, the doctor gently presses PAMS into the patient's back to create skin indentations demarcating the needle insertion point. These indentations are not affected by skin sterilisation, and may improve accuracy and reduce the time taken to perform the epidural procedure. Next, the angle between the ultrasound probe and the patient's back can be measured using PAMS, and this angle can be maintained using a needle guide during the epidural procedure.

The purpose of this randomised study is to evaluate the usability of PAMS and to identify areas for further improvement.

This study will involve up to 10 healthy simulated patients, and up to 30 volunteer ultrasound operators. After undergoing a standardised training session with a mannequin, the ultrasound operators will be randomly assigned to perform skin marking on the simulated patients as though they are performing an ultrasound-guided epidural anaesthesia procedure (no needle puncture will be made) using either PAMS, or standard clinical practice with marker pens. After completing the procedure, the ultrasound operators will cross over and perform the procedure again using either PAMS or standard clinical practice with marker pens.

Both the ultrasound operators and simulated patients will be asked to complete satisfaction and usability surveys regarding their experience with the procedures.

DETAILED DESCRIPTION:
The volunteer ultrasound operators are women's anaesthesiologists trained in the use of ultrasound-guided neuraxial procedures.

Simulated patients are healthy volunteers from other departments, without spine abnormalities.

The ultrasound operators will be asked to complete a questionnaire regarding your prior experience with neuraxial ultrasonography and undergo structured training on the use of PAMS using a mannequin. Next, they will be asked to perform the following two procedures (the order at which they will perform the procedures will be randomised):

1. Ultrasound scan using PAMS

   * After attaching PAMS to the ultrasound probe, they will perform a lumbar ultrasound scan on a simulated patient to identify the desired needle insertion site and gently press PAMS into the simulated patient's back to create skin indentations demarcating the desired needle insertion site.
   * Next, adjust the angulation of the ultrasound probe to optimise the image of the simulated patient's lumbar spine, and read the angle between the ultrasound probe and patient's back off a graduated scale.
   * Remove the ultrasound probe, and position the needle-insertion guide corresponding to the skin indentations. Needle angulation can be simulated by mounting a blunt needle on to the insertion guide.
   * Finally, they will be asked to complete a usability questionnaire.
2. Ultrasound scan without PAMS (standard clinical practice)

   * Perform a lumbar ultrasound scan to identify the desired needle insertion site, followed by demarcation using skin markers.
   * Next, adjust the angulation of the ultrasound probe to optimise the image of the simulated patient's lumbar spine.
   * Remove the ultrasound probe and simulate needle insertion by touching the tip of a blunt needle to the patient's back, at the desired angle.
   * Finally, they will then be asked to complete a usability questionnaire.

Both procedures are non-invasive (i.e. no skin punctures will be made). No follow up is required for this study.

No new research medications are involved in this study.

Additionally, video recordings may be made of the procedures. Any video or ultrasound images obtained during the course of this study will be stored and analysed only for the purposes of this study for a period not exceeding 7 years, and will be destroyed after completion of the study. Technical data such as the scanning duration and success rate will also be documented.

ELIGIBILITY:
Ultrasound operators

Inclusion Criteria:

* Anaesthesiologists
* Trained in the use of ultrasound-guided neuraxial procedures

Exclusion Criteria:

* No experience with ultrasound-guided neuraxial procedures

Simulated patients

Inclusion Criteria:

* Healthy, no significant medical comorbidity (American Society of Anesthesiologists Physical Status I or II)
* No spinal abnormalities, or previous spinal surgery

Exclusion Criteria:

* Significant spinal abnormality
* Previous spinal surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2021-08-31 (Estimated); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
Satisfaction survey of simulated patients and operators | Immediately after performing the procedure
  Satisfaction and feedback regarding the respective procedures

SECONDARY OUTCOMES:
Time taken to perform procedure | Immediately after performing the procedure
  Comparison of time taken to perform the interventional procedure (PAMS), versus standard clinical practice (control)

CONTACTS AND LOCATIONS:
Locations (1):
- KK Women's and Children's Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tan HS, Sng BL, Sia ATH. Reducing breakthrough pain during labour epidural analgesia: an update. Curr Opin Anaesthesiol. 2019 Jun;32(3):307-314. doi: 10.1097/ACO.0000000000000713. PMID 31045638